CLINICAL TRIAL: NCT01437553
Title: Registry Using IVUS and iMAP to Evaluate Atherosclerotic Coronary Plaque in Acute Coronary Syndromes
Brief Title: Imaging Whole Coronary Artery With Intravascular Ultrasound (Ivus) And Imap For Plaque Tissue Composition In Patients With Acute Myocardial Infarction
Acronym: iWONDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Cristiano Freitas de Souza, M.D., Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BSCI-01
Record Dates: First submitted 2011-09-18; First posted 2011-09-21 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Acute Coronary Syndrome
Keywords: IVUS; iMAP; Catheterization; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVUS (Other): Patients undergoing catheterization due to acute coronary syndrome will have IVUS done with grayscale and iMAP analysis performed.
  Interventions: Device: iMAP

INTERVENTIONS:
Device: iMAP — IVUS and iMAP analysis for acute coronary syndromes

SUMMARY:
The iWONDER trial has the following objective:

To analyze the morphological, phenotypic and tissue characteristics of atherosclerotic plaques angiographically considered "culprit" and "not-culprit" in patients undergoing coronary angiography due to STEMI (ST-elevation myocardial infarction).

DETAILED DESCRIPTION:
Coronary artery angiography (CA) is a two-dimensional silhouette of the arterial lumen from a complex three dimensional vascular structure. This exam has several limitations already well documented, including shortening of the vessel, overlapping images, intra and inter-observer variability during the consideration of the severity of injuries. Besides, it offers great limitations in the diagnosis of the composition of atherosclerotic plaque. Furthermore, intravascular ultrasound (IVUS) provides a sensitive and reproducible measure of the dimensions of the vessel and allows direct visualization of the vessel wall, atherosclerotic plaque and arterial lumen. The utility of grayscale IVUS as prognostic tool and as a guide in percutaneous coronary interventions (PCI) is well established. More recently, IVUS has also provided new insights for safety and efficacy of drug eluting stent (DES).

Advances in technology now allow IVUS to characterize the morphology and composition of plaques. Specifically, the analysis of the IVUS wave frequency - beyond the interpretation of wave lengths used in grayscale IVUS- enables in vivo analysis of atherosclerotic plaque composition with high sensitivity and specificity. Although previous studies have reported data using IVUS radiofrequency analysis, the use of a new modality (iMapTM, Boston Scientific, Santa Clara, CA, USA) for characterization of atherosclerotic plaque is poorly known.

ELIGIBILITY:
Inclusion Criteria:

* Age < 75 years
* Diagnosis of NSTEMI/STEMI with prior use of fibrinolytics in the past 7 days
* Signature of the Term of Informed Consent

Exclusion Criteria:

* Hemodynamic instability
* Clinical signs of post-AMI ventricular dysfunction (Killip III/IV)
* Angiographic findings of (1)coronary anatomy with significant tortuosity, (2) critical coronary obstruction preventing the passage of the IVUS catheter and (3) total occlusion of any of the three epicardial coronary arteries.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Atherosclerotic plaque composition | Patients will be followed during in-hospital period, an expect average of 7 days
  Atherosclerotic plaque composition of "culprit" and "non-culprit" lesions will be evaluated using grayscale IVUS and iMAP analysis in patients presenting with acute coronary syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano M Caixeta, PhD, Principal Investigator — Federal University of São Paulo; Cristiano F Souza, MD, Principal Investigator — Federal University of São Paulo; Antonio C Carvalho, PhD, Study Director — Federal University of São Paulo; Claudia M Alves, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil